CLINICAL TRIAL: NCT01175902
Title: To Prove the Non-inferiority of Cosopt Compared to Xalatan in the Aspects of Intraocular Pressure and Ocular Perfusion Pressure in Subjects With Normal Tension Glaucoma
Brief Title: Intraocular Pressure and Ocular Perfusion Pressure of Cosopt in Normal Tension Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Chan Kee Park, Seoul St. Mary's Hospital, The Catholic University of Korea
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: cosopt-IOP/OPP
Record Dates: First submitted 2010-07-26; First posted 2010-08-05 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2014-12

CONDITIONS: Normal Tension Glaucoma
Keywords: Normal tension glaucoma
MeSH Terms: conditions — Low Tension Glaucoma | interventions — dorzolamide-timolol combination; Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Latanoprost first, then Dorzolamide/Timolol Patients first on Latanoprost eyedrops once a day, then on Dorzolamide/Timolol twice a day
  Interventions: Drug: dorzolamide/timolol; Drug: latanoprost
- Arm 2 (Active Comparator): Dorzolamide/Timolol first, then Latanoprost Patients first on Dorzolamide/Timolol eyedrops twice a day, then on Latanoprost eyedrops once a day
  Interventions: Drug: dorzolamide/timolol; Drug: latanoprost

INTERVENTIONS:
Drug: dorzolamide/timolol — dorzolamide/timolol fixed combination eyedrop, 2 times a day
  Other Names: Cosopt
Drug: latanoprost — compare with dorzolamide/timolol fixed combination eyedrop one time a day
  Other Names: Xalatan

SUMMARY:
To prove the non-inferiority of the fixed timolol-dorzolamide combination (Cosopt) compared to 0.005% latanoprost (Xalatan) in the aspects of intraocular pressure (IOP) and ocular perfusion pressure (OPP) in subjects with normal tension glaucoma (NTG)

Clinical hypotheses. Primary hypothesis

* Cosopt group is non-inferior to Xalatan group in diurnal IOP reduction.

Secondary hypothesis

* Cosopt group is non-inferior to Xalatan group in diurnal diastolic and systolic OPP.

DETAILED DESCRIPTION:
Cosopt (dorzolamide/timolol fixed combination) has well known effect for IOP reduction in POAG and OHT.3-5 However, there is no study about the effect and safety of Cosopt in NTG, Cosopt is not used the first line drug in the management of NTG.

In Korea, the prevalence of NTG is higher than western countries, the majority (about 80-90%) of open angle glaucoma patients have an IOP of 21 mmHg or less, so the study of NTG is important and searching of effective drug for the treatment of NTG is necessary.

In this study, we would prove the non-inferiority of Cosopt compared to Xalatan,6 which is used as a first line drug in the management of NTG, in the aspects of IOP and OPP including diastolic OPP (DOPP).

A prospective, interventional, randomized, crossover, single masked, single center study. Forty-four NTG patients were randomly allocated to one of two groups. Patients in group A were treated with Cosopt, lubricant, and Xalatan for 4 weeks each, whereas patients in group B were treated with Xalatan, lubricant, and Cosopt for 4 weeks each.

Recruit NTG patients, who are not treated with the glaucoma medication recent 2 months. If treated, after washout period of 4 weeks, the patients can be included in the study. Baseline IOP, systolic and diastolic BP will be measured. (Day 1) After 4 weeks of treatment of Cosopt or Xalatan, all participants will be checked diurnal IOP, systolic and diastolic BP. IOP was measured by Goldmann applanation tonometry (mean of three consecutive readings) with the patient in a sitting position at the slit lamp. Every IOP will be measured by one masked glaucoma specialist who is unaware of the treatment assignments. After the IOP measurements, after a 5-minite rest, pulse rate and BP (systolic and diastolic) of radial artery were measured in the sitting position using a standard automated blood pressure cuff. During the period, all measuring instruments keep to be calibrated by the manufacturer's instruction.

- OPP was calculated according to the following formula: OPP=(1/3 systolic BP + 2/3 diastolic BP) x 2/3 -IOP, diastolic OPP (DOPP)=diastolic BP-IOP. During the 4 weeks washout period, subjects will use lubricants.(Week 8) In this crossover study, with the other eye drops, the same measurement will be performed. (Week 12)

ELIGIBILITY:
The identification of NTG was based on reproducible glaucomatous visual field defects, corresponding to typical ONH changes.

Unilateral or bilateral visual field loss (description as below) as determined by at least two consecutive automated static threshold perimetry tests.

One eye is randomly selected in the cases where both eyes are treated.

Inclusion criteria:

1. age ranging from 45 to 75 years
2. best-corrected visual acuity no worse than 20/30 Snellen equivalent
3. optic nerve head cupping (i.e., a vertical cup-to-disc ratio of more than 0.6) and/or notching of neuroretinal rim, and/or retinal nerve fiber defects characteristic of glaucoma
4. visual field loss (i.e., a localized defect with at least three adjacent nonedge points depressed >5 dB from the normal value, and a nucleus of at least one point depressed 10 dB from the normal value)
5. repeated measurements of untreated IOP, which documented values less than 22 mmHg
6. central corneal thickness ranging from 540 to 560 microns
7. open-angle confirmed by gonioscopy

Exclusion criteria:

1. active or chronic systemic diseases and/or concomitant assumption of any medication known to affect IOP, BP and/or HR
2. corneal abnormalities preventing reliable applanation tonometry
3. severe ocular trauma, ocular inflammation or infection, intraocular surgery or argon laser treatment or laser trabeculoplasty
4. myopic or other fundus changes preventing reliable optic disc evaluation,
5. visual field defects caused by nonglaucomatous disease
6. history of allergy to the ingredients of Cosopt or Xalatan eye drops

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chan Kee Park, M.D., PhD., Principal Investigator — The Catholic University of Korea
Locations (1):
- Seoul St. Mary's hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee NY, Park HY, Park CK. Comparison of the Effects of Dorzolamide/Timolol Fixed Combination versus Latanoprost on Intraocular Pressure and Ocular Perfusion Pressure in Patients with Normal-Tension Glaucoma: A Randomized, Crossover Clinical Trial. PLoS One. 2016 Jan 12;11(1):e0146680. doi: 10.1371/journal.pone.0146680. eCollection 2016. PMID 26756747

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seoul St. Mary's Hospital From April, 5th, 2011 to October, 16th, 2014
Pre-assignment Details: 44 enrolled, 44 completed
Groups:
- Latanoprost: Patients on Latanoprost eyedrops
  dorzolamide/timolol fixed combination: Cosopt eyedrop, 2 times a day
  latanoprost: compare with Cosopt one time a day
- Dorzolamide/Timolol: Patients on Dorzolamide/Timolol eyedrops
  dorzolamide/timolol fixed combination: Cosopt eyedrop, 2 times a day
  latanoprost: compare with Cosopt one time a day
Period: Overall Study
Arm/Group | Latanoprost | Dorzolamide/Timolol
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Latanoprost | Dorzolamide/Timolol | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.72 (7.42) | 59.68 (7.12) | 60.20 (7.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 22 | 22 | 44
Spherical equivalent [Mean (Standard Deviation); unit: diopters] — Sperical equvalaent comes from refractive error of the patient and it is calcaulated as the algebraic sum of the value of the sphere and half the cylindrical value.
  diopters | -0.74 (1.95) | -1.04 (2.71) | -0.89 (2.34)
Central corneal thickness [Mean (Standard Deviation); unit: micrometers] | 542.73 (11.43) | 544.23 (17.33) | 543.48 (14.53)
Mean deviation of visual field [Mean (Standard Deviation); unit: decibels] | -4.00 (3.79) | -2.92 (2.96) | -3.46 (3.41)

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP), Period 1
Description: IOP (mean IOP) after 4 weeks of treatment
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Latanoprost, Period 1: Patients on Latanoprost eyedrops
  dorzolamide/timolol fixed combination: Cosopt eyedrop, 2 times a day
  latanoprost: compare with Cosopt one time a day
- Dorzolamide/Timolol, Period 1: Patients on Dorzolamide/Timolol eyedrops
  dorzolamide/timolol fixed combination: Cosopt eyedrop, 2 times a day
  latanoprost: compare with Cosopt one time a day
Arm/Group | Latanoprost, Period 1 | Dorzolamide/Timolol, Period 1
Number analyzed (Participants) | 22 | 22
mmHg
  IOP at 8am | 13.72 (2.93) | 13.50 (3.09)
  IOP at 10am | 13.27 (2.37) | 13.36 (2.75)
  IOP at 12pm | 13.54 (2.30) | 12.63 (2.98)
  IOP at 16pm | 13.77 (2.50) | 13.77 (2.61)
  IOP at 20pm | 13.36 (1.89) | 13.63 (2.46)
Statistical Analysis 1: Comparison: Latanoprost, Period 1 vs Dorzolamide/Timolol, Period 1; Comparison between two arms were made for IOP, systolic BP, diastolic BP and OPP at each time period; Test type: Non-Inferiority or Equivalence — To prove the non-inferiority of Cosopt to Xalatan, the sample size calculation was based on the assumption that non-inferiority margin of trough IOP of 1.5mmHg. A sample size of n=21 patients per group, this study has 80% power (1-β=0.80) and α=0.05, crossover-designed analysis. In this study, the upper limit of the 95% CI is expected above the maximal acceptable clinically significant difference of 1.5 mmHg of IOP; p = 0.05, t-test, 2 sided — Comparison between two arms were made for IOP, systolic BP, diastolic BP and OPP at each time period; Comparison between two arms were made for IOP, systolic BP, diastolic BP and OPP at each time period; Mean Difference (Final Values) = 0.9 — Comparison between two arms were made for IOP, systolic BP, diastolic BP and OPP at each time period

2. Primary Outcome: Intraocular Pressure (IOP), Period 2
Description: IOP (mean IOP) after treaemt from week 8 to week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Latanoprost, Period 2: Patients on Latanoprost eyedrops
  dorzolamide/timolol fixed combination: Cosopt eyedrop, 2 times a day
  latanoprost: compare with Cosopt one time a day
- Dorzolamide/Timolol, Period 2: Patients on Dorzolamide/Timolol eyedrops
  dorzolamide/timolol fixed combination: Cosopt eyedrop, 2 times a day
  latanoprost: compare with Cosopt one time a day
Arm/Group | Latanoprost, Period 2 | Dorzolamide/Timolol, Period 2
Number analyzed (Participants) | 22 | 22
mmHg
  IOP at 8am | 13.13 (3.02) | 12.36 (2.51)
  IOP at 10am | 12.81 (3.21) | 12.36 (2.55)
  IOP at 12pm | 12.54 (3.05) | 12.72 (2.45)
  IOP at 16pm | 12.81 (3.24) | 13.04 (2.41)
  IOP at 20pm | 13.40 (2.36) | 13.13 (2.07)

3. Primary Outcome: Blood Pressure (BP), Period 1
Description: systolic and diastolic BP at 4 weeks after use of eyedrops
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Latanoprost, Period 1 | Dorzolamide/Timolol, Period 1
Number analyzed (Participants) | 22 | 22
mmHg
  systolic BP at 8am | 121.82 (16.25) | 122.82 (17.90)
  systolic BP at 10am | 120.68 (12.76) | 119.14 (18.01)
  systolic BP at 12pm | 120.45 (13.22) | 120.55 (17.23)
  systolic BP at 16pm | 122.09 (13.14) | 118.55 (18.74)
  systolic BP at 20pm | 123.32 (14.09) | 119.45 (18.92)
  diastolic BP at 8am | 74.77 (11.45) | 77.36 (8.59)
  diastolic BP at 10am | 74.50 (11.13) | 73.81 (7.32)
  diastolic BP at 12pm | 74.22 (9.71) | 73.18 (7.53)
  diastolic BP at 16pm | 75.27 (10.35) | 72.81 (6.94)
  diastolic BP at 20pm | 75.95 (11.78) | 74.13 (7.52)

4. Primary Outcome: Blood Pressure (BP), Period 2
Description: systolic and diastolic BP measured after treaemt from week 8 to week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Latanoprost, Period 2 | Dorzolamide/Timolol, Period 2
Number analyzed (Participants) | 22 | 22
mmHg
  systolic BP at 8am | 123.14 (12.58) | 118.41 (15.47)
  systolic BP at 10am | 123.59 (12.06) | 117.95 (12.73)
  systolic BP at 12pm | 122.41 (11.89) | 119.05 (13.999)
  systolic BP at 16pm | 124.50 (12.78) | 118.45 (14.90)
  systolic BP at 20pm | 123.23 (14.88) | 119.82 (13.34)
  diastolic BP at 8am | 76.45 (7.71) | 73.72 (9.67)
  diastolic BP at 10am | 74.86 (8.40) | 72.50 (7.70)
  diastolic BP at 12pm | 75.54 (7.89) | 72.40 (8.39)
  diastolic BP at 16pm | 73.45 (7.50) | 71.36 (8.78)
  diastolic BP at 20pm | 73.81 (8.64) | 74.72 (7.32)

5. Secondary Outcome: Ocular Perfusion Pressure (OPP), Period 1
Description: OPP was calculated according to the following formula:
  OPP=(1/3 systolic BP + 2/3 diastolic BP) x 2/3 -IOP, diastolic OPP (DOPP)=diastolic BP-IOP
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Latanoprost, Period 1 | Dorzolamide/Timolol, Period 1
Number analyzed (Participants) | 22 | 22
mmHg
  OPP at 8am | 46.57 (8.34) | 49.12 (6.76)
  OPP at 10am | 46.65 (6.81) | 46.95 (6.06)
  OPP at 12pm | 46.21 (6.64) | 48.17 (5.51)
  OPP at 16pm | 46.81 (7.14) | 45.44 (5.98)
  OPP at 20pm | 47.79 (7.34) | 46.73 (6.73)

6. Secondary Outcome: OPP, Period 2
Description: OPP was calculated according to the following formula:
  OPP=(1/3 systolic BP + 2/3 diastolic BP) x 2/3 -IOP, diastolic OPP (DOPP)=diastolic BP-IOP
  OPP after treaemt from week 8 to week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Latanoprost, Period 2 | Dorzolamide/Timolol, Period 2
Number analyzed (Participants) | 22 | 22
mmHg
  OPP at 8am | 48.36 (6.00) | 46.71 (7.34)
  OPP at 10am | 48.04 (5.98) | 46.07 (5.96)
  OPP at 12pm | 48.47 (5.98) | 45.90 (6.00)
  OPP at 16pm | 47.81 (6.21) | 44.99 (5.80)
  OPP at 20pm | 47.10 (6.70) | 46.70 (5.14)

ADVERSE EVENTS:
Time Frame: During the 12 weeks study period
Arm/Group | Latanoprost | Dorzolamide/Timolol
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No